CLINICAL TRIAL: NCT07396597
Title: Investigation of Respiratory Functions, Muscle Strength, Physical Activity Level, and Quality of Life in Individuals With Premature Ventricular Complexes
Brief Title: Physical Impairments in Premature Ventricular Complex
Status: Not yet recruiting | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Gulsah Bargi, Principal Investigator, Izmir Democracy University
Other Study IDs: Premature Ventricular Complex
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Premature Ventricular Complexes
Keywords: cough; muscle strength; quality of life; pulmonary function; ventricular premature complexes,
MeSH Terms: conditions — Ventricular Premature Complexes; Cough | interventions — Polyvinyl Chloride

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ventricular premature complexes group: This group will consist of individuals with premature ventricular complex.
  Interventions: Other: Physical Evaluations of Patients with Premature Ventricular Complex
- Control Group: This group will consist of healthy individuals.
  Interventions: Other: Physical Evaluations of Healthy Individuals

INTERVENTIONS:
Other: Physical Evaluations of Patients with Premature Ventricular Complex — In this study, data from individuals with premature ventricular complex will be collected through face-to-face assessments. Respiratory functions, respiratory and peripheral muscle strength, cough strength, physical activity level, and quality of life will be assessed in these individuals who meet the inclusion criteria. All data obtained through these assessments will be collected from participants face-to-face at one time and for a maximum of approximately 1 hour.
  Groups: Ventricular premature complexes group
Other: Physical Evaluations of Healthy Individuals — In this study, data from healthy individuals will be collected through face-to-face assessments. Respiratory functions, respiratory and peripheral muscle strength, cough strength, physical activity level, and quality of life will be assessed in these individuals who meet the inclusion criteria.All data obtained through these assessments will be collected from participants face-to-face at one time and for a maximum of approximately 1 hour.
  Groups: Control Group

SUMMARY:
Premature ventricular complexes may be observed in individuals without underlying disease due to factors such as physical inactivity, advanced age, smoking, male sex, and psychosocial disturbances, and in some cases may result in sudden cardiac death. Therefore, the aim of this study is to investigate respiratory function, respiratory muscle strength, cough strength, handgrip strength, physical activity level, and quality of life in individuals with premature ventricular complexes.

DETAILED DESCRIPTION:
The primary aim of this study is to comprehensively investigate respiratory function, respiratory muscle strength, cough strength, handgrip strength, physical activity level, and quality of life in individuals with premature ventricular complexes. Additionally, an important secondary aim is to identify potential differences in these parameters between individuals with premature ventricular complexes and healthy controls and to contribute original findings to the existing literature.Participants will be evaluated in terms of these parameters through clinical assessments, questionnaires, and measurements.

ELIGIBILITY:
Inclusion Criteria for Individuals with Premature Ventricular Complexes (PVCs):

* Aged between 18 and 80 years
* Presence of symptomatic premature ventricular complexes resistant to ≥1 antiarrhythmic medication (including β-blockers and calcium channel blockers)
* Premature ventricular complex burden ≥10%
* Ventricular arrhythmias originating from any focus (or foci) within the right or left ventricle
* Physically able to participate in all study assessments
* Willingness to participate in the study by providing written informed consent

Inclusion Criteria for Control Group Participants:

* Aged between 18 and 80 years
* Healthy individuals
* Willingness to participate in the study
* Physically able to participate in all study assessments

Exclusion Criteria for Individuals with Premature Ventricular Complexes (PVCs):

* Left ventricular ejection fraction (LVEF) <45% unless PVC-induced cardiomyopathy is documented (defined as a >15% improvement in LVEF following reduction of PVC burden through pharmacological therapy or ablation)
* Progressive decline in LVEF within the last 4 months, regardless of etiology
* Severe heart failure classified as New York Heart Association (NYHA) Class ≥III
* Ventricular arrhythmias attributed to underlying structural heart disease, known myocardial scar, or myocarditis
* Change in the dosage of antiarrhythmic medications (including β-blockers and calcium channel blockers) within 2 months prior to enrollment
* Failed catheter ablation within 3 months prior to enrollment
* Known thyroid disorders or individuals undergoing renal dialysis
* Life expectancy <12 months
* Presence of angina pectoris
* Diagnosis of chronic obstructive pulmonary disease (COPD) or asthma
* Resting heart rate >120 beats/min
* Resting systolic blood pressure ≥180 mmHg
* Resting diastolic blood pressure ≥100 mmHg
* Resting peripheral oxygen saturation ≤90%

Exclusion Criteria for Control Group Participants:

* Presence of premature ventricular complexes
* Presence of any acute or chronic medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults including individuals diagnosed with symptomatic premature ventricular complexes and healthy control participants. Participants will be recruited from patients presenting to the Cardiology Department of Buca Seyfi Demirsoy Training and Research Hospital and volunteers without premature ventricular complexes.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Maximal inspiratory pressure (MIP) | through study completion, an average of 1 year
  The MIP which shows respiratory muscle strength will be evaluated using a portable mouth pressure measuring device based on American Thoracic Society and European Respiratory Society criteria.

SECONDARY OUTCOMES:
Maximal expiratory pressure (MEP) | through study completion, an average of 1 year
  The MEP which shows respiratory muscle strength will be evaluated using a portable mouth pressure measuring device based on American Thoracic Society and European Respiratory Society criteria.
Forced vital capacity (FVC) | through study completion, an average of 1 year
  Pulmonary function (Forced vital capacity (FVC)) will be evaluated with a spirometer.
Forced expiratory volume in the first second (FEV1) | through study completion, an average of 1 year
  Pulmonary function (Forced expiratory volume in the first second (FEV1)) will be evaluated with a spirometer.
FEV1 / FVC | through study completion, an average of 1 year
  Pulmonary function (FEV1 / FVC) will be evaluated with a spirometer.
Peak flow rate (PEF) | through study completion, an average of 1 year
  Pulmonary function (Peak flow rate (PEF)) will be evaluated with a spirometer.
Cough Strength | through study completion, an average of 1 year
  Participants' peak cough expiratory flow (PCEF) values will be assessed in an upright sitting position using a peak cough flow meter (ExpiRite Peak Flow Meter, China). Following a deep inspiration, participants will be instructed to cough as forcefully as possible into the device. The best value obtained from at least three trials will be recorded.
Handgrip Strength | through study completion, an average of 1 year
  Maximum isometric strength of the hand and forearm muscles will be measured using a hydraulic hand dynamometer.Measurements will be performed in an upright sitting position in accordance with guidelines. The mean of the three measurements for the right and left hands will be used for analysis.
Assessment of Physical Activity | through study completion, an average of 1 year
  Participants' physical activity levels over the previous seven days will be assessed using the International Physical Activity Questionnaire-Short Form. The questionnaire consists of 7 items that assess time spent walking, and moderate- and vigorous-intensity physical activities over the last seven days. Total physical activity scores will be calculated by summing the duration (minutes) and frequency (days) of walking, moderate-intensity, and vigorous-intensity activities. Total physical activity score will be expressed as metabolic equivalent task minutes per week (MET-min/week).
Assessment of Quality of Life | through study completion, an average of 1 year
  Participants' quality of life will be evaluated using the Short Form-36 Health Survey. The SF-36 assesses eight health domains: general health, physical functioning, role limitations due to physical problems, role limitations due to emotional problems, social functioning, bodily pain, vitality, and mental health, along with one additional item assessing health transition. Participants will be instructed to respond to each question in a manner that best reflects their current condition, and researchers will provide clarifying guidance when necessary.

CONTACTS AND LOCATIONS:
Overall Officials: GÜLŞAH BARĞI, Study Director — Izmir Democracy University; ESRA SUDE AKIN, Principal Investigator — Izmir Democracy University; DEFNE FİL, Principal Investigator — Izmir Democracy University; ERKAN ALPASLAN, Principal Investigator — Izmir Democracy University
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeppenfeld K, Tfelt-Hansen J, de Riva M, Winkel BG, Behr ER, Blom NA, Charron P, Corrado D, Dagres N, de Chillou C, Eckardt L, Friede T, Haugaa KH, Hocini M, Lambiase PD, Marijon E, Merino JL, Peichl P, Priori SG, Reichlin T, Schulz-Menger J, Sticherling C, Tzeis S, Verstrael A, Volterrani M; ESC Scientific Document Group. 2022 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death. Eur Heart J. 2022 Oct 21;43(40):3997-4126. doi: 10.1093/eurheartj/ehac262. No abstract available. PMID 36017572
- [Background] Aktan R, Ocaker Aktan O, Ozalevli S, Dursun H. Impact of Inspiratory Muscle Strength and Lung Function on Functional Exercise Capacity in Post-myocardial Infarction Patients: A Cross-sectional Study. Thorac Res Pract. 2025 Oct 24;26(6):307-313. doi: 10.4274/ThoracResPract.2025.2025-7-5. Epub 2025 Sep 18. PMID 40960384